CLINICAL TRIAL: NCT05269329
Title: Double-blind Placebo-controlled Multicenter Randomized Clinical Trial to Assess Efficacy and Safety of HC8, Film-coated Tablets, 10 mg (Valenta Pharm, Russia) in Patients With Dry Non-productive Cough Against Acute Respiratory Viral Infection
Brief Title: Efficacy and Safety of XC8, Film-coated Tablets, 10 mg in Patients With Dry Non-productive Cough Against Acute Respiratory Viral Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC8-02-01-2020
Record Dates: First submitted 2022-01-28; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: Common Cold; Acute Respiratory Infection; Influenza, Human
MeSH Terms: conditions — Common Cold; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- XC8, film-coated tablets, 20 mg/day (Experimental)
  Interventions: Drug: XC8, film-coated tablets, 20 mg/day
- XC8, film-coated tablets, 40 mg/day (Experimental)
  Interventions: Drug: XC8, film-coated tablets, 40 mg/day
- XC8, film-coated tablets, 80 mg/day (Experimental)
  Interventions: Drug: XC8, film-coated tablets, 80 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC8, film-coated tablets, 20 mg/day — 20 mg/day (1 tablet twice a day)
  Arms: XC8, film-coated tablets, 20 mg/day
Drug: XC8, film-coated tablets, 40 mg/day — 40 mg/day (2 tablets twice a day)
  Arms: XC8, film-coated tablets, 40 mg/day
Drug: XC8, film-coated tablets, 80 mg/day — 80 mg/day (4 tablets twice a day)
  Arms: XC8, film-coated tablets, 80 mg/day
Drug: Placebo — 1, 2, or 4 tablets twice a day
  Arms: Placebo

SUMMARY:
Study to assess the efficacy and safety of XC8, film-coated tablets, 10 mg in comparison with placebo in patients with dry non-productive cough against acute respiratory infections, and to determine the dosing regimen of XC8, film-coated tablets, 10 mg for treatment of dry non-productive cough against acute respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

1. Signing and dating of the IPP informed consent form by the patient.
2. Women and men between the ages of 18 and 65 years, inclusive, at the time of signing the informed consent form.
3. Clinical diagnosis of acute respiratory viral infection of the upper respiratory tract (ICD-10 code J00-J06) or acute bronchitis (J20, J21 according to ICD-10).
4. Onset of disease symptoms no more than 3 days prior to screening.
5. Presence of a patient with a dry unproductive cough.
6. Frequency of cough episodes ≥10 in the past 24 h before the screening visit and randomization.
7. Cough frequency rated by the patient as 3-4 on the daytime cough section and 2-4 on the nighttime cough section of the Daytime and Nighttime Cough Scales.
8. Patient rating of cough severity on the DRS ≥ 4 points.
9. No indication for therapy due to BHSA infection at the time of study inclusion: negative rapid test for Group A β-haemolytic streptococcus.
10. For women of preserved reproductive potential, a negative pregnancy test and agreement to use approved contraceptive methods for the duration of study participation, beginning at visit 0, and for 3 weeks after the end of the study; for men, agreement to use approved contraceptive methods throughout the study participation period and for 3 weeks after the end of the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the active ingredient or any of the excipients of the study drug/placebo.
2. Known or suspected hypersensitivity to acetylcysteine.
3. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
4. Trauma (including open wounds in the mouth and erosive-desquamous lesions of the oral mucosa) and/or oropharyngeal burns, scarlet fever, rubella, measles, mumps at the time of screening or within 3 months prior to screening.
5. Acute obstructive laryngitis or suspected obstructive laryngitis.
6. Presence of signs of laryngeal stenosis (stridor, shortness of breath).
7. Exacerbation of chronic bronchitis or chronic obstructive pulmonary disease (COPD).
8. Bronchial asthma, including a history.
9. History of tuberculosis.
10. History of pulmonary emphysema.
11. Acute or chronic pneumonia, or suspected pneumonia.
12. Condition after intubation.
13. Gastroesophageal reflux being the primary cause of cough (as judged by the investigating physician).
14. Allergic rhinitis as primary cause of cough (according to study physician).
15. Body temperature > 39.0 °C.
16. Presence of at least one of the epidemic signs: return from a foreign trip 14 days prior to the onset of symptoms; presence of close contact in the past 14 days with a person under COVID-19 surveillance who has subsequently become ill; having close contact in the past 14 days with a person who has a laboratory-confirmed diagnosis of COVID-19; having occupational contacts with an individual with a suspected or confirmed case of COVID-19.
17. Positive result of laboratory testing for SARS-CoV-2 RNA using nucleic acid amplification techniques or SARS-CoV-2 antigen using immunochromatographic analysis at the time of screening.
18. The need for systemic antibiotic therapy and/or other drugs/procedures from the list of prohibited therapies/procedures.
19. Use of analgesics or antipyretics within 12 hours prior to screening.
20. Use of glucocorticosteroids, β-adrenoblockers, ACE inhibitors, theophylline drugs, expectorants, cough suppressants, anesthetics, anti-allergic drugs (leukotriene receptor antagonists, H1-histamine receptor blockers, sodium cromoglycate preparations), antiviral drugs, immunosuppressants, systemic antibacterial drugs for 7 days before screening.
21. History of smoking more than 10 pack/years (pack-years: number of cigarettes smoked per day multiplied by the number of years of smoking divided by 20).
22. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels ≥ 2.5 × highest normal value, serum bilirubin levels ≥ 1.5 × highest normal value.
23. Glomerular filtration rate (GFR) ≤ 60 ml/min.
24. History of cancer of the respiratory system.
25. History of other malignancies, except for patients who have not had the disease in the past 5 years, patients with fully cured basal cell carcinoma of the skin, or fully cured carcinoma in situ.
26. Serious cardiovascular disease at the time of screening or within 12 months prior to screening, including: New York Heart Association Class III or IV chronic heart failure, severe arrhythmias requiring treatment with antiarrhythmic drugs, unstable angina pectoris, myocardial infarction, heart and coronary artery surgery, transient ischemic attack or stroke, uncontrolled hypertension with systolic blood pressure > 180 mm Hg Std. and diastolic blood pressure >110 mmHg, pulmonary embolism.
27. Other severe, decompensated or unstable somatic diseases (any disease or condition that threatens the patient's life or worsens the patient's prognosis, or makes it impossible for the patient to participate in a clinical trial).
28. Patient's unwillingness or inability to comply with protocol procedures (in the opinion of the research physician).
29. Pregnancy or breastfeeding (for women).
30. Alcoholism, drug dependence, substance abuse history and/or at the time of screening.
31. A history of schizophrenia, schizoaffective disorder, bipolar disorder or other psychiatric pathology.
32. Participation in another clinical trial within 3 months prior to inclusion in the study.
33. Other conditions that, in the opinion of the investigating physician, preclude inclusion of the patient in the study.

Withdrawal Criteria:

1. Identification of a probable or confirmed case of COVID-19
2. Ineffectiveness of therapy - persistence or increased frequency of cough attacks ≥ 1 by visit 3 (day 8-9) compared to visit 1 (day 1).
3. AEs requiring withdrawal of study drug/placebo.
4. The occurrence of any disease or condition during the study that, in the opinion of the study physician, worsens the patient's prognosis and also makes it impossible for the patient to continue participating in the clinical trial.
5. Erroneous inclusion of a patient who does not meet the inclusion criteria and/or meets the inclusion criteria.
6. Taking any of the drugs of prohibited therapy, performing a prohibited procedure.
7. The necessity of prescribing prohibited concomitant therapy/procedures.
8. Pregnancy of the patient.
9. Patient's desire to stop participating in the study.
10. Lack of adequate cooperation of the patient with the doctor-researcher during the study.
11. Other protocol violations that are significant in the opinion of the physician-researcher.
12. Other administrative reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Coughing frequency | The estimate will include data from 24 hours to Day 1 and Day 5
  Change in coughing frequency by ≥ -50% by day 5 relative to visit 1

SECONDARY OUTCOMES:
Frequency of cough episodes | The assessment will include data for 24 h before days 5, 8, 11, and 15, respectively.
  Frequency of cough episodes by 5, 8, 11, and 15 days after visit 1
Time to clinical cough cure | From Day 1 (visit 1) to the first day of consecutive days on which ≤ 1 point on the Daytime Cough and Nighttime Cough Scales sections of the Daytime and Nighttime Cough Scales is recorded, assessed up to Day 16 (visit 5).
  Time (days) from visit 1 to achievement of clinical cough cure. Clinical cough cure is defined as having ≤ 1 score on the Daytime Cough and Nighttime Cough Scales for at least 3 consecutive days.
Proportion of patients with ≤ 1 score on the daytime cough and nighttime cough Scales sections | The daytime cough section score will include data for days 4, 7, 10, and 14, respectively. The nighttime cough section score will include data for the night preceding days 5, 8, 11, and 15, respectively.
  Proportion of patients with ≤ 1 score on the daytime cough and nighttime cough Scales sections by days 5, 8, 11, and 15 after visit 1.
Change (score) in cough severity | The score will include data 24 h before days 5, 8, 11, and 15, respectively.
  Change (score) in cough severity according to the digital rating scale (DRS) by days 5, 8, 11, and 15 compared to visit 1.
Time (days) from visit 1 to a reduction in cough severity | From Day 1 (visit 1) up to Day 16 (visit 5).
  Time (days) from visit 1 to a reduction in cough severity by DRS of ≥2 points.
Percentage of patients prescribed acetylcysteine | From Day 1 (visit 1) up to Day 16 (visit 5).
  Percentage of patients who were prescribed acetylcysteine for the conversion of dry to wet cough.
Time (days) from visit 1 to administration of acetylcysteine | From Day 1 (visit 1) up to Day 16 (visit 5).
  Estimated only in patients who were prescribed acetylcysteine.
Proportion of patients dropped out of the study due to prescription of systemic antibiotic therapy. | From Day 1 (visit 1) up to Day 16 (visit 5).
  Proportion of patients dropped out of the study due to prescription of systemic antibiotic therapy due to the development of complications of the disease
Time (days) from visit 1 to achieving ≤ 1 score on the daytime cough | From Day 1 (visit 1) up to Day 16 (visit 5).
  Time (days) from visit 1 to achieving ≤ 1 score on the daytime cough section Scales of daytime and nighttime cough.
Change (score) in daytime cough | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Change (score) in daytime cough section Daytime and nighttime cough scales (from 0 - no cough episodes to 5 - severe cough, which makes normal activity impossible) by days 4, 7, 10, and 14 compared to visit 1.
Proportion of patients with a score ≤ 1 on the daytime cough | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Proportion of patients with a score ≤ 1 on the daytime cough section Daytime and nighttime cough scales by days 4, 7, 10, and 14 after visit 1.
Percentage of patients with ≥1 point decrease in daytime cough | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Percentage of patients with ≥1 point decrease in daytime cough section Daytime and nighttime cough scales by 4, 7, 10, and 14 days post-visit 1.
Proportion of patients with ≥ 2 points reduction in daytime cough | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Proportion of patients with ≥ 2 points reduction in "daytime cough" Scales of daytime and nighttime cough by 4, 7, 10, and 14 days after visit 1.
Time (days) from visit 1 to reaching ≤ 1 score on the nighttime cough | From Day 1 (visit 1) up to Day 16 (visit 5).
  Time (days) from visit 1 to reaching ≤ 1 score on the nighttime cough section Scales for daytime and nighttime cough.
Change (score) in the nighttime cough | Assessment will include data for the night before days 5, 8, 11, and 15, respectively.
  Change (score) in the nighttime cough section Day and night cough scales (from 0 - no cough episodes to 5 - cough that prevents a subject from falling asleep) by days 5, 8, 11, and 15 compared to visit 1.
Proportion of patients with a score ≤ 1 on nighttime cough | Assessment will include data for the night before days 5, 8, 11, and 15, respectively.
  Proportion of patients with a score ≤ 1 on nighttime cough Scales of day and night cough by days 5, 8, 11, and 15 after visit 1.
Percentage of patients with ≥1 point decrease in nighttime cough | Assessment will include data for the night before days 5, 8, 11, and 15, respectively.
  Percentage of patients with ≥1 point decrease in nighttime cough section Scales of day and night cough by 5, 8, 11, and 15 days after visit 1.
Percentage of patients with a reduction of ≥ 2 points in the nighttime cough | Assessment will include data for the night before days 5, 8, 11, and 15, respectively.
  Percentage of patients with a reduction of ≥ 2 points in the nighttime cough section Day and night cough scales by days 5, 8, 11, and 15 after visit 1.
Change in the number of episodes of nocturnal awakening due to cough | Assessment will include data for the night before days 5, 8, 11, and 15, respectively.
  Change in the number of episodes of nocturnal awakening due to cough by days 5, 8, 11, and 15 compared to visit 1.
Time (days) to attain ≤ 1 score for each symptom | From Day 1 (visit 1) up to Day 16 (visit 5).
  Time (days) to attain ≤ 1 score for each symptom on the Acute Respiratory Infection Major Symptom Rating Scale
Proportion of patients with attainment of ≤ 1 point on each symptom | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Proportion of patients with attainment of ≤ 1 point on each symptom on the Acute Respiratory Infection Major Symptom Rating Scale by days 4, 7, 10, and 14
Percentage of patients with a decrease of ≥1 score on each symptom | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Percentage of patients with a decrease of ≥1 score on each symptom on the Acute Respiratory Infection Major Symptom Rating Scale by days 4, 7, 10, and 14
Change in each symptom score | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Change in each symptom score on the Acute Respiratory Infection Major Symptom Rating Scale by days 4, 7, 10, and 14 compared to visit 1.
Proportion of patients with body temperature ≤ 37.0 °C | From Day 3-4 (visit 2) up to Day 16 (visit 5).
  Proportion of patients with body temperature ≤ 37.0 °C by Visits 2-5. Patients who had a body temperature ≤ 37.0°C at Visit 1 will not be included in the analysis for that symptom.
Percentage of patients with complete resolution of all symptoms | Assessment will include data for days 4, 7, 10, and 14, respectively.
  Percentage of patients with complete resolution of all acute respiratory infection symptoms by days 4, 7, 10, and 14.
Proportion of patients with "very high" and "high" efficacy | From Day 3-4 (visit 2) up to Day 16 (visit 5).
  Proportion of patients with "very high" and "high" efficacy at visits 2, 3, 4, and 5 by physician's assessment.
Proportion of patients with each category of Global Assessment scale | From Day 3-4 (visit 2) up to Day 16 (visit 5).
  Proportion of patients with each category of Global Assessment by the physician at visits 2, 3, 4, and 5.
Safety - Adverse Events (AEs) | From visit 0 up to Day 20 +/- 2 (visit 6).
  Total number of AEs stratified by severity and frequency
Safety - Adverse Reactions | From visit 0 up to Day 20 +/- 2 (visit 6).
  Frequency of Adverse Reactions
Safety - Serious adverse events (SAEs) | From visit 0 up to Day 20 +/- 2 (visit 6).
  Frequency of SAEs associated with the use of the study drug/placebo
Safety - Percentage of patients with at least one AE | From visit 0 up to Day 20 +/- 2 (visit 6).
  Percentage of patients with at least one AE
Safety - Percentage of patients who interrupted the treatment due to AE | From visit 0 up to Day 20 +/- 2 (visit 6).
  Percentage of patients who interrupted the treatment due to the occurrence of AE

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Ivanovo Kuvaev Clinical Hospital, Ivanovo
  - Kirov State Medical University, Kirov
  - Unimed-C Jsc, Moscow
  - Professors' Clinic LLC., Perm
  - EosMED JSC, Saint Petersburg
  - Aurora MedFort LLC, Saint Petersburg
  - Private Healthcare Institution Clinical Hospital "RZD-Medicine" of St. Petersburg, Saint Petersburg
  - OrKli Hospital LLC., Saint Petersburg
  - Medical Diagnostic Center LLC., Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided